CLINICAL TRIAL: NCT04906785
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-385 High-dose in Healthy Volunteers Under Fed Conditions
Brief Title: Clinical Study to Investigate the PK Profiles and Safety of CKD-385 in Healthy Volunteers Under Fed Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A88_11BE2110
Record Dates: First submitted 2021-05-27; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence1 (Experimental): 1. Period 1: Reference drug(D744)
  2. Period 2: Test drug(CKD-385)
  Interventions: Drug: CKD-385; Drug: D744
- Sequence2 (Experimental): 1. Period 1: Test drug(CKD-385)
  2. Period 2: Reference drug(D744)
  Interventions: Drug: CKD-385; Drug: D744

INTERVENTIONS:
Drug: CKD-385 — Test Drug
Drug: D744 — Reference Drug

SUMMARY:
Clinical Study to Investigate the PK Profiles and Safety of CKD-385 in Healthy Volunteers Under Fed Conditions

DETAILED DESCRIPTION:
A randomized, open-label, single dose, crossover study to evaluate the pharmacokinetic profiles and safety of CKD-385 high-dose in healthy volunteers under fed conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults age≥19 years and age<55 years at the time of screening
2. Individuals who had 17.5 kg/m2 ≤ Body Mass Index(BMI) < 30.5kg/m2 and men's total body weight ≥ 55 kg, women's total body weight ≥ 45 kg

   * BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years
4. Individuals who were deemed to be appropriate as study subjects following laboratory tests (hematology, blood chemistry, urinalysis, viral/ bacterial, etc.) and vital signs, ECG etc. performed at screening
5. Individuals who signed an informed consent form approved by the IRB of Chonbuk National University Hospital and decided to participate in the study after being fully informed of the study prior to participation, including the objective, content and characteristics of the investigational product
6. Individuals who agreed proper contraception during the study and did consent to not donation of sperm 1 month after the last dose of study drug infusion
7. Individuals with the ability and willingness to participate the entire study period

Exclusion Criteria:

1. Subject who has (or has histories of) clinically significant blood, kidney, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, liver, mental, neurological or allergic diseases(except for asymptomatic seasonal allergy at the time of administration) or evidence(except for simple dental history such as dental calculus, impacted tooth, wisdom tooth, etc.)
2. Subject with a history of gastrointestinal disorders(esophageal achalasia or esophagus stenosis, Crohn's disease) or gastrointestinal surgery(except for simple appendicitis surgery or hernia surgery or tooth extraction surgery) that may affect the absorption of drug
3. Subject who shows the following values as a result of laboratory tests

   *ALT or AST > 2 times upper limit of normal range
4. Subject who has a history of regular alcohol consumption in excess of 210 g/week within 6 months of screening
5. Subject who smokes more than one pack of cigarette a day within 6 months of screening
6. Subject who took other clinical trial drugs or bioequivalence test drugs within 3 months before the first administration of clinical trial drug
7. Subject who conform to the specific items below

   * systolic blood pressure less than 90 mmHg, greater than 140 mmHg or diastolic blood pressure less than 60 mmHg or greater than 90 mmHg in a sitting position
   * Severe bradycardia (less than 50 beats/minute)
8. Subject who has significant alcohol abuse or drug abuse within a year of screening
9. Subject who took drugs which are known as disturbing drug metabolism within 30 days prior to the first administration of clinical trial drug.
10. Subject who uses any of other drugs, including over-the-counter medications and prescription medications within 10 days prior to first administration of clinical trial drug.
11. Subject who donated whole blood within 2 months prior to first administration of clinical trial drug or blood components within 1 month prior to first administration of clinical trial drug
12. Subject who is hypersensitive to the components of a clinical trial drug or clinical trial drug itself.
13. Subject had genetic dysfunctions like galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
14. Subject who is not able to consume high-fat meal provided during the clinical trial
15. Subjects who were deemed inappropriate to participate in the study by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-06-04 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-08-06 (Estimated)

PRIMARY OUTCOMES:
AUCt of CKD-385 | Pre-dose (0 hour), 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Area under the concentration-time curve from time zero to time of CKD-385

SECONDARY OUTCOMES:
AUCinf of CKD-385 | Pre-dose (0 hour), 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Area under the concentration-time curve from zero up to infinity of CKD-385
Tmax of CKD-385 | Pre-dose (0 hour), 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Time to maximum plasma concentration of CKD-385
T1/2 of CKD-385 | Pre-dose (0 hour), 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Terminal elimination half-life of CKD-385
CL/F of CKD-385 | Pre-dose (0 hour), 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Apparent clearance of CKD-385
Vd/F of CKD-385 | Pre-dose (0 hour), 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Apparent Volume of Distribution of CKD-385

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No